CLINICAL TRIAL: NCT03482297
Title: Randomized, Double-blind, Sham-controlled to Evaluate the Effects of an Automated Abdominal Binder in Improving Orthostatic Tolerance in Autonomic Failure Patients With Disabling Orthostatic Hypotension
Brief Title: Automated Abdominal Binder for Orthostatic Hypotension
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Luis E Okamoto, Research Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 151008; 1R01HL144568-01A1 (NIH)
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Orthostatic Hypotension; Autonomic Failure; Pure Autonomic Failure; Multiple System Atrophy
Keywords: orthostatic hypotension; abdominal binder; pure autonomic failure; multiple system atrophy
MeSH Terms: conditions — Hypotension, Orthostatic; Pure Autonomic Failure; Multiple System Atrophy | interventions — Midodrine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, sham-controlled, parallel-group, 3-study days inpatient study to compare the efficacy of the automated abdominal binder versus sham treatment in improving orthostatic tolerance in patients with primary autonomic failure disabled by neurogenic orthostatic hypotension.
Who Masked: Participant, Investigator
Masking Description: Patients and investigators will be blinded as to the experimental interventions (active or sham abdominal binder, and placebo or midodrine pills)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Automated Abdominal Binder (Experimental): Participants will be studied on three separate study days, two days apart: one day for baseline measurements (placebo pill t.i.d), one day for treatment with 10 mg midodrine t.i.d (standard of care), and one day for treatment with the automated abdominal binder combined with placebo pill t.i.d The automated abdominal binder will be placed during the morning orthostatic trial on the active/sham binder study day. The binder will inflate automatically (~40 mmHg) every time the participant stands up throughout the study day.
  Interventions: Device: automated abdominal binder; Drug: Placebo; Drug: Midodrine
- Sham binder (Sham Comparator): Participants will be studied on three separate study days, two days apart: one day for baseline measurements (placebo pill t.i.d), one day for treatment with 10 mg midodrine t.i.d (standard of care), and one day for treatment with the sham binder combined with placebo pill t.i.d. The sham binder will be placed during the morning orthostatic trial on the active/sham binder study day. The sham binder will inflate automatically (~5 mmHg) every time the participant stands up throughout the study day.
  Interventions: Device: Sham binder; Drug: Placebo; Drug: Midodrine

INTERVENTIONS:
Device: automated abdominal binder — The binder automatically inflates every time the participant stands up to apply a compression level of about 40 mmHg. Participants will wear the device throughout the active/sham study day.
  Arms: Automated Abdominal Binder
Device: Sham binder — The binder automatically inflates every time the participant stands up to apply a compression level of about 5 mmHg. Participants will wear the device throughout the active/sham study day.
  Arms: Sham binder
Drug: Placebo — Oral placebo will be given three times a day on the baseline day (placebo)
Drug: Midodrine — A midodrine pill 10mg will be given three times a day on the standard of care study day

SUMMARY:
The automated inflatable abdominal binder is an investigational device for the treatment of orthostatic hypotension (low blood pressure on standing) in patients with autonomic failure. The purpose of this study is to determine safety and effectiveness of the automated abdominal binder in improving orthostatic tolerance in these patients.

DETAILED DESCRIPTION:
This is a randomized, double-blind, sham-controlled, parallel group study to compare the efficacy of the automated abdominal binder (inflated to 40 mm Hg) versus sham treatment (abdominal binder inflated to 5 mm Hg) in improving orthostatic tolerance in patients with primary autonomic failure disabled by orthostatic hypotension.

Potential participants will be admitted to the Vanderbilt Clinical Research Center for evaluation of inclusion and exclusion criteria. Eligible patients will be randomized to the active or sham binder group. Patients will then be asked to participate on three separate study days, two days apart: one day for baseline measurements (placebo pill t.i.d), one day for treatment with 10 mg midodrine t.i.d (standard of care), and one day for treatment with active or sham binder combined with placebo pill t.i.d. The order of the study days will be randomized. On each study day, blood pressure and heart rate will be measured while sitting, lying down, standing and walking during the Morning Orthostatic Trial, and posture and walking tests.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 40-80 years.
* Possible or probable Multiple Systems Atrophy and Pure Autonomic Failure as defined by Consensus Criteria.
* Neurogenic orthostatic hypotension defined as a ≥30-mm Hg decrease in SBP within 3 minutes of standing associated with impaired autonomic reflexes determined by autonomic testing in the absence of other identifiable causes, and
* Moderate to severe orthostatic symptoms, defined as an Orthostatic Hypotension Symptom Assessment (OHSA) composite score ≥4 (self-rating Likert scale of 0 to 10, with 0 reflecting absence of symptoms), within the first 10 minutes of the screening orthostatic stress test, and that have an impact in quality of life, as defined by the patient.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy.
* Systemic illnesses known to produce autonomic neuropathy, including but not limited to diabetes mellitus, amyloidosis, monoclonal gammopathies, and autoimmune neuropathies.
* History of known aortic aneurisms, thoracic, abdominal or pelvic surgery in the past 6 months; symptomatic abdominal or inguinal hernias; severe gastroesophageal reflux; recent fractures or fissures of ribs, thoracic or lumbar spine; medical devices implanted on the abdominal wall or abdomen that would interfere with the binder; known abdominal or pelvic tumors, cysts or enlarged spleen; intolerance to any increase in intraabdominal pressure.
* Pre-existing sustained supine hypertension ≥180/110.
* Bedridden patients or those who are unable to stand due to motor impairment or severe orthostatic hypotension.
* Clinically unstable coronary artery disease (recurrent angina despite medical therapy), or major cardiovascular or neurological event in the past 6 months (myocardial infarction, stroke or transient ischemic attacks).
* Concomitant use of anticoagulants

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Orthostatic tolerance | After 10 minutes of standing (or as tolerated) during the Morning orthostatic trial on the automated binder/sham study day
  orthostatic tolerance is defined as the area under the curve of the upright systolic blood pressure (AUCSBP) during the Morning Orthostatic Trials
Orthostatic Hypotension Symptom Assessment (OHSA) Score | After 10 minutes of standing (or as tolerated) during the Morning orthostatic trial on the automated binder/sham study day
  The Orthostatic Hypotension Symptom Assessment (OHSA) Score is the part I of the Orthostatic Hypotension Questionnaire (OHQ). It consists of six questions, each rating the intensity of one characteristic symptom of orthostatic hypotension: 1. Dizziness, lightheadedness, feeling faint, or feeling like you might black out; 2. Problems with vision (blurring, seeing spots, tunnel vision, etc.); 3. Generalized weakness; 4. Fatigue; 5. Trouble concentrating; and 6. Head/neck discomfort.The items are scored on an 11-point Likert scale from 0 to 10, with 0 indicating no symptoms and 10 indicating the worst possible symptoms. Composite score is the average of the item scores obtained at the post-intervention stand period during the Morning Orthostatic Trials

SECONDARY OUTCOMES:
Upright time | After 10 minutes of standing and 15 minutes waking (as tolerated)
  Sum of standing and walking times

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Professor of Medicine and Pharmacology; Luis E Okamoto, MD, Principal Investigator — Research Assistant Professor
Locations (1):
- Autonomic Dysfunction Center/ Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No